CLINICAL TRIAL: NCT06908941
Title: The Cardiovascular Benefits of Dark Chocolate Supplementation Before High-intensity Resistance Exercise in the Early Follicular and Mid-luteal Phases of the Menstrual Cycle
Brief Title: The Cardiovascular Benefits of Resistance Training and Dark Chocolate in Female Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Cheng-Shiun He, PhD, Professor, National Cheng Kung University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CCUREC111122101
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Vascular Function in Healthy Volunteers
Keywords: dark chocolate; estrogen; cardiovascular function

STUDY DESIGN:
Intervention Model Description: EF-MC: early follicular-milk chocolate EF-DC: early follicular-dark chocolate ML-MC: Mid Luteal-milk chocolate ML-DC: Mid Luteal-dark chocolate
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Follicular (Experimental): Participants consumed either 85% dark chocolate or milk chocolate (1g/kg body weight) before high-intensity resistance exercise during the early follicular (days 2-5) phases of two menstrual cycles.
  Interventions: Dietary Supplement: dark chocolate; Dietary Supplement: milk chocolate; Behavioral: high-intensity resistance exercise
- Mid-Luteal (Active Comparator): Participants consumed either 85% dark chocolate or milk chocolate (1g/kg body weight) before high-intensity resistance exercise during the mid-luteal (days 18-24) phases of two menstrual cycles.
  Interventions: Dietary Supplement: dark chocolate; Dietary Supplement: milk chocolate; Behavioral: high-intensity resistance exercise

INTERVENTIONS:
Dietary Supplement: dark chocolate — Participants consumed 85% dark chocolate (1g/kg body weight) before high-intensity resistance exercise during the early follicular (days 2-5) and mid-luteal (days 18-24) phases of two menstrual cycles. Finger-toe pulse wave velocity (ftPWV), arterial stiffness, blood pressure, and plasma NO levels were measured at rest, 2 hours after chocolate consumption (baseline), immediately post-exercise (T0), and at 60 (T60) and 120 (T120) minutes post-exercise.
Dietary Supplement: milk chocolate — Participants consumed milk chocolate (1g/kg body weight) before high-intensity resistance exercise during the early follicular (days 2-5) and mid-luteal (days 18-24) phases of two menstrual cycles. Finger-toe pulse wave velocity (ftPWV), arterial stiffness, blood pressure, and plasma NO levels were measured at rest, 2 hours after chocolate consumption (baseline), immediately post-exercise (T0), and at 60 (T60) and 120 (T120) minutes post-exercise.
Behavioral: high-intensity resistance exercise — Participants performed high-intensity resistance exercise during the early follicular (days 2-5) and mid-luteal (days 18-24) phases of two menstrual cycles.

SUMMARY:
This study investigates the effects of 85% dark chocolate supplementation on vascular function and nitric oxide (NO) levels during high-intensity resistance exercise in healthy women across menstrual phases. Using a randomized crossover design, 31 women consumed either dark chocolate or milk chocolate before exercising during the early follicular and mid-luteal phases. Vascular markers, including pulse wave velocity (ftPWV), arterial stiffness, blood pressure, and plasma NO levels, were measured at multiple time points.

DETAILED DESCRIPTION:
Background:

Dark chocolate, rich in flavanols, may support vascular health by reducing arterial stiffness and blood pressure across menstrual phases. This study examined the effects of 85% dark chocolate on nitric oxide (NO) levels and vascular function during high-intensity resistance exercise in healthy women across the early follicular and mid-luteal phases.

Methods:

Thirty-one healthy women (aged 20-30 years) with regular menstrual cycles completed a randomized, crossover study (conducted at National Chung Cheng University, Sep-Dec 2023). Participants consumed either 85% dark chocolate or milk chocolate (1g/kg body weight) before high-intensity resistance exercise during the early follicular (days 2-5) and mid-luteal (days 18-24) phases of two menstrual cycles. Finger-toe pulse wave velocity (ftPWV), arterial stiffness, blood pressure, and plasma NO levels were measured at rest, 2 hours after chocolate consumption (baseline), immediately post-exercise (T0), and at 60 (T60) and 120 (T120) minutes post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* the healthy adult women,
* aged 20-30 years, from a local university campus,
* had a regular menstrual cycles in the past three months.

Exclusion Criteria:

* (1) irregular menstrual cycles (menstrual cycle length < 21 or > 35 days in the past three months),
* (2) pregnancy or lactation in the past year,
* (3) history of cardiovascular or uterine surgery in the past six months,
* (4) use of contraceptives or other female hormone medications,
* (5) smoking or alcohol consumption habits,
* (6) hypertension (blood pressure > 140/90 mmHg), chronic diseases, heart disease, or other cardiovascular conditions, (7) allergy to cocoa products, nuts, or fruits.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Finger-Toe Pulse Wave Velocity (ftPWV) | Finger-toe pulse wave velocity (ftPWV) were measured at rest, 2 hours after chocolate consumption (baseline), immediately post-exercise (T0), and at 60 (T60) and 120 (T120) minutes post-exercise.
  Measurements at other time points are taken while participants are resting in the laboratory. Firstly, sensors for photoplethysmography (PPG) were placed on the right index finger and right big toe of the participants. These sensors were marked with an oily pen to ensure consistent placement throughout the experiment. The signals were then amplified using a Biopec MP150 (MP150, Biopac Systems Inc., Goleta, CA, USA), with each physiological signal collected for at least 150 seconds. The signals were analyzed using MATLAB to calculate the time difference between the two pulse waves. The length of the participant's body segments ( sternum to the right index finger, and sternum to the big toe of the right foot) was measured, and this value was divided by the average difference between 10 pulse waves (in the stable interval of 150 seconds) to calculate the ftPWV value (m/s).

SECONDARY OUTCOMES:
Arterial Index | Arterial index (API and AVI) were measured at rest, 2 hours after chocolate consumption (baseline), immediately post-exercise (T0), and at 60 (T60) and 120 (T120) minutes post-exercise.
  The arterial pressure volume index (API) and arterial velocity pulse index (AVI) are measured using the PASESA AVE-2000 (PASESA, Tokyo, Japan) with a wrapped around the right upper arm of seated participants. The API reflected the stiffness of peripheral arteries by assessing the pressure-volume relationship of the artery, while the AVI primarily reflected the stiffness of central arteries by analyzing the ratio of forward and reflected pressure waves. Each measurement was taken three times, and the average of the three readings was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Shiun He Professor, Principal Investigator — National Chung Cheng University
Locations (1):
- National Chung Cheng University, Chiayi County, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaynor-Metzinger SHA, Triplett NT, Meucci M, Fasczewski KS, Flinchum DH, Collier SR. Central arterial stiffness, wave reflection, and heart rate variability following 4-week high-intensity resistance training intervention in young active women. Eur J Appl Physiol. 2022 Oct;122(10):2283-2293. doi: 10.1007/s00421-022-05003-4. Epub 2022 Jul 19. PMID 35852625
- [Derived] Wang CW, Fang SH, Yu TA, Chen LY, Wang CK, Wang SC, He CS. The Cardiovascular Benefits of Dark Chocolate Supplementation before High-Intensity Resistance Exercise in the Early Follicular and Mid-Luteal Phases of the Menstrual Cycle. Sports Med Open. 2025 Apr 18;11(1):39. doi: 10.1186/s40798-025-00850-9. PMID 40249472
- See also: National Chung Cheng University Human Research Ethics Center — https://rec.ccu.edu.tw/p/412-1152-3134.php?Lang=zh-tw
- Available data/document: Informed Consent Form: CCUREC111122101 — https://rec.ccu.edu.tw/p/412-1152-3134.php?Lang=zh-tw — National Chung Cheng University Human Research Ethics Center